CLINICAL TRIAL: NCT01708616
Title: A Single-center, Randomized, Double-blind, Two-period Crossover Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of the Combination of Multiple Doses of RO5285119 With a Single Dose of Risperidone in Healthy Subjects
Brief Title: A Study of the Combination of Multiple Doses of RO5285119 With a Single Dose of Risperidone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Double
Other Study IDs: BP28318; 2012-003231-31 (EudraCT Number)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo + risperidone (Placebo Comparator)
  Interventions: Drug: RO5285119 placebo; Drug: risperidone
- Placebo +placebo (Placebo Comparator)
  Interventions: Drug: RO5285119 placebo; Drug: risperidone placebo
- RO5285119 + placebo (Active Comparator)
  Interventions: Drug: RO5285119; Drug: risperidone placebo
- RO5285119 + risperidone (Experimental)
  Interventions: Drug: RO5285119; Drug: risperidone

INTERVENTIONS:
Drug: RO5285119 — multiple doses
  Arms: RO5285119 + placebo; RO5285119 + risperidone
Drug: RO5285119 placebo — multiple doses
  Arms: Placebo + risperidone; Placebo +placebo
Drug: risperidone — single dose
  Arms: Placebo + risperidone; RO5285119 + risperidone
Drug: risperidone placebo — single dose
  Arms: Placebo +placebo; RO5285119 + placebo

SUMMARY:
This single-center, randomized, double-blind, two-period crossover study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic effects of the combination of multiple doses of RO5285119 with a single dose of risperidone in healthy volunteers. Subjects will be randomized to one of 4 treatment sequences of two periods to receive multiple doses of RO5285119 plus a single dose of risperidone or risperidone placebo or multiple doses of RO5285119 placebo plus a single dose of risperidone or risperidone placebo, with a washout period of approximately 3 weeks between treatment periods. Anticipated time on study is up to 12 weeks (from screening through study completion).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, 18 - 50 years of age inclusive Healthy status is defined by absence of evidence of any active or chronic disease following detailed medical and surgical history and a physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Women have to be postmenopausal or surgically sterile
* Male subjects must use a barrier method of contraception for the duration of the study and for 3 months after last dosing

Exclusion Criteria:

* Suspicion of regular consumption of drug of abuse, or history of drug or alcohol abuse
* Positive for hepatitis B, hepatitis C or HIV infection
* History of clinically significant hypersensitivity or allergic reactions
* Disorders of the central nervous system, including psychiatric disorders, behavioural disturbances, cerebrovascular events, depression, bipolar disorder, migraine, Parkinson
* Regular smoker (>5 cigarettes, >3 pipe-fulls, >3 cigars per day)
* Administration of an investigational drug or device within 3 months prior to first dosing

  * Hypersensitivity to risperidone or any of its excipients
* Any other known contraindications to risperidone as stated in the SmPC

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single dose risperidone in combination with multiple doses of RO5285119: Maximum plasma concentration (Cmax) | Pre-dose to 24 hours post-dose
Pharmacokinetics of single dose risperidone in combination with multiple doses of RO5285119: Area under the concentration-time curve (AUC) | Pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 12 weeks
Pharmacodynamic markers for risperidone: Prolactin levels | Pre-dose to 6 hours post-dose
Pharmacodynamic assessments for risperidone: Level of sedation | Pre-dose to 24 hours post-dose
Pharmacokinetics of RO5285119 in combination with single dose risperidone: Maximum plasma concentration (Cmax) | Day 1 to Day 18
Pharmacokinetics of RO5285119 in combination with single dose risperidone: Area under the concentration-time curve (AUC) | Day1 to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France